CLINICAL TRIAL: NCT04784130
Title: Enhancing Diabetes and Hypertension Self-Management for Rural Appalachian Patients In Patient-Centered Medical Homes
Brief Title: Enhancing Diabetes and Hypertension Self-Management Rural Appalachian Patients In Patient-Centered Medical Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Ranjita Misra, Professor, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1908672206
Record Dates: First submitted 2020-07-29; First posted 2021-03-05 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Diabetes Mellitus, Type 2; Hypertension
Keywords: diabetes; hypertension; self-management
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Diabetes Mellitus | interventions — Exercise; Diet Therapy

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DHSMP core (Experimental): Dietary Modification and Physical Activity
  Interventions: Behavioral: Physical Activity; Behavioral: Dietary Modification
- DHSMP core plus (Experimental): Dietary Modification, physical activity and medication adherence
  Interventions: Behavioral: Physical Activity; Behavioral: Medication Adherence; Behavioral: Dietary Modification
- DHSMP control (Active Comparator): enhanced usual care-3 hours of education plus materials.
  Interventions: Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Physical Activity — Respondents will complete activity logs (step count, using pedometer) and surveys (two items from the Summary of Diabetes Self-care activities measure) for physical activity.
Behavioral: Medication Adherence — Respondents will provide information on their medication adherence using a survey (questionnaire - MMAS-8).
  Arms: DHSMP core plus
Behavioral: Dietary Modification — Respondents will complete food logs and surveys (three items from the Summary of Diabetes Self-care activities measure) for dietary intake.
  Arms: DHSMP core; DHSMP core plus

SUMMARY:
The goal of this R34 planning project is to test the feasibility and acceptability of a 12-week modified diabetes and hypertension self-management program using trained Health Coaches.

DETAILED DESCRIPTION:
West Virginians have one of the highest prevalence of comorbid diabetes and hypertension in the nation that pose an enormous disease and economic burden in this medically underserved state. Self-management of these two commonly found chronic conditions are an essential component of comprehensive disease management. The goal of this R34 planning project is to test the feasibility and acceptability of a 12-week culturally-tailored, multimodal, diabetes and hypertension self-management program with a core (diet and physical activity) versus core plus (diet, physical activity and medication adherence) to an enhanced usual care (EUC) control group. Seventy-five eligible adults with comorbid diabetes and hypertension will be randomized with a 1:1:1 ratio, based on allocation sequence generated by the bio-statistician investigator in the team. The study will examine the extent to which key components (diet, physical activity, and medication adherence) contribute to the differences in clinical outcomes (HbA1c and blood pressure) between three groups using quantitative and qualitative focus groups and the RE-AIM evaluation framework. The longer term effects of the intervention will be evaluated in a subsequent R01 clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* English speaking adults ≥ 18 years of age;
* co-occurring diagnosis of type 2 diabetes and hypertension
* body mass index ≥ 25.0
* willing to be randomized, and complete the intervention and all assessments.

Exclusion Criteria:

* currently pregnant or breastfeeding
* diagnosed with a severe mental illness
* have any condition that requires physical activity limitations or is contraindicated for the Dietary Assessment to Stop Hypertension (DASH) diet
* inability to complete the study protocol.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Clinical outcomes-BP | 6 months after enrollment
  Difference in BP between baseline and end of program
Clinical Outcomes-A1c | 6 months after enrollment
  Difference in A1c between baseline and end of program

SECONDARY OUTCOMES:
Behavioral outcome - dietary modification for high fat foods; question | 6 months after enrollment
  Dietary analysis will be based on consumption of high fat foods (such as red meat or full-fat dairy) at baseline and completion of the Program. All participants will be assessed regarding the number of days they eat high fat foods using a survey question from the Summary of Diabetes Self-care activities measure by Toolbert et al., Diabetes Care, 2000. "On how many of the last SEVEN DAYS did you eat high fat foods such as red meat or full-fat dairy products?" 0 1 2 3 4 5 6 7. Changes in mean number of days of eating high fat foods will be assessed at baseline and at the completion of the program.
Behavioral outcome - healthy eating plan; questions | 6 months after enrollment
  Dietary analysis will be based on following a healthy eating plan at baseline and completion of the Program. All participants will be assessed regarding the number of days they followed a healthful eating plan using a survey question from the Summary of Diabetes Self-care activities measure by Toolbert et al., Diabetes Care, 2000. "How many of the last SEVEN DAYS have you followed a healthful eating plan?" 0 1 2 3 4 5 6 7. Changes in mean number of days followed a healthy eating plan will be assessed at baseline and at the completion of the program.
Behavioral outcome - dietary modification for fruits and vegetables; questions | 6 months after enrollment
  Dietary analysis will be based on eating fruits and vegetables at baseline and completion of the Program. All participants will be assessed regarding the number of days they eat five or more servings of fruits and vegetables using a survey question from the Summary of Diabetes Self-care activities measure by Toolbert et al., Diabetes Care, 2000. "On how many of the last SEVEN DAYS did you eat five or more servings of fruits and vegetables?" 0 1 2 3 4 5 6 7. Changes in mean number of days of eating fruits and vegetables will be assessed at baseline and at the completion of the program.
Behavioral outcome - Activity log; Step count, using pedometer | 6 months after enrollment
  All participants will be asked to wear a pedometer to record their daily step count.
Behavioral outcome - exercise; questions | 6 months after enrollment
  All participants will be assessed regarding the number of days they exercise using two survey questions from the Summary of Diabetes Self-care activities measure by Toolbert et al., Diabetes Care, 2000. The description of the questions are as follow: Q1. "On how many of the last SEVEN DAYS did you participate in at least 30 minutes of physical activity? (please list the total minutes of continuous activity, including walking)" 0 1 2 3 4 5 6 7 & Q2. "On how many of the last SEVEN DAYS did you participate in a specific exercise session (such as swimming, walking, biking) other than what you do around the house or as part of your work?" 0 1 2 3 4 5 6 7). The total exercise score will be calculated by the mean number of days for the two questions). Changes in mean number of days exercised will be assessed at baseline and at the completion of the program.
Behavioral outcome - medication adherence; questions | 6 months after enrollment
  Respondents will provide information on their medication adherence using a survey (questionnaire - MMAS-8). Changes in medication adherence will be assessed at baseline and completion of the program.

CONTACTS AND LOCATIONS:
Locations (1):
- Clark K. Sleeth Family Medicine Center, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No